CLINICAL TRIAL: NCT00190944
Title: Effects of Teriparatide on Distal Radius Fracture Healing
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8175; B3D-MC-GHCN
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-10-12 (Estimated); Status verified 2007-10

CONDITIONS: Colles' Fracture
MeSH Terms: conditions — Colles' Fracture | interventions — Teriparatide

INTERVENTIONS:
Drug: Teriparatide
Drug: placebo

SUMMARY:
Effects of Teriparatide on Distal Radius Fracture Healing

ELIGIBILITY:
Inclusion Criteria:

Ambulatory, postmenopausal, women 45 to 85 years of age. Postmenopausal is defined as at least 2 years without regular menses

Sustained a unilateral, dorsally angulated fracture of the distal radius within 10 days

Received conservative treatment of her distal radius fracture, including closed reduction and immobilization device (such as cast, splint, or brace)

Free of severe or chronically disabling conditions other than a distal radius fracture as determined by the investigator

Without language barrier, cooperative, expected to return for all follow-up procedures, and has given informed consent before entering the study and after being informed of the risks, medications and procedures to be used in the study.

In the opinion of the investigator, the patient is willing to be trained and use the pen-injector daily, is able to satisfactorily use a pen-type injection delivery system, or is willing to receive daily subcutaneous injections from a care partner who has been trained to use the pen injector

Exclusion Criteria:

Increased baseline risk of osteosarcoma

History of a malignant neoplasm in the 5 years prior to visit 2, with the exception of superficial basal cell carcinoma or squamous cell carcinoma of the skin that has been definitely treated

Have currently known, suspected, or history of other diseases that affect bone metabolism other than postmenopausal osteoporosis or cause secondary osteoporosis that has been clinically active in the 1 year prior to visit 2

Have elevated serum calcium values

Active liver disease or clinical jaundice

History of symptomatic nephro-or urolithiasis in the 2 years prior to visit 2

Previous fractures or bone surgery in the currently fractured distal forearm

Joint disease such as rheumatoid arthritis or disabling osteoarthritis that clearly affect the function of the wrist and/or hand of the injured arm

Requirement for chronic treatment with nonsteroidal anti-inflammatory drugs defined as more than 3 consecutive months of any NSAID treatment

Treatment with:

Oral bisphosphonates for more than 18 months during the prior 3 years, or have received any oral or intravenous biphosphonate therapy within the last 2 months prior to screening.

Oral strontium ranelate for any duration

Systemic corticosteroids for more than 30 days (total) in the 6 months prior to visit 2, or any systemic corticosteroid dose in the 1 month prior to visit 2. Ophthalmic, oric, topical, or nasally inhaled corticosteroid therapy may be used without these restrictions.

Fluoride at therapeutic doses (greater than or equal to 20mg/day) for more than 3 months during the last 2 years or for more than a total of 2 years, or any dosages within the 6 months prior to visit 2.

Ages: 45 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105
Dates: Start 2004-12; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Time to radiographic healing

SECONDARY OUTCOMES:
There are no secondary outcomes for this trial

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST, Study Director — Eli Lilly and Company
Locations (7):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New York, New York, United States
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterrey, Mexico
- Poland (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lublin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
- Romania (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucharest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Timișoara
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Linköping, Sweden

REFERENCES:
- [Derived] Aspenberg P, Genant HK, Johansson T, Nino AJ, See K, Krohn K, Garcia-Hernandez PA, Recknor CP, Einhorn TA, Dalsky GP, Mitlak BH, Fierlinger A, Lakshmanan MC. Teriparatide for acceleration of fracture repair in humans: a prospective, randomized, double-blind study of 102 postmenopausal women with distal radial fractures. J Bone Miner Res. 2010 Feb;25(2):404-14. doi: 10.1359/jbmr.090731. PMID 19594305
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com